CLINICAL TRIAL: NCT00933452
Title: A Open Single-dose and Multiple-dose Study to Evaluate the Pharmacokinetics and Safety of Duloxetine in Chinese Han Healthy Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics of Duloxetine in Chinese Han Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Jiangsu Nhwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: LI, Huafang, Shanghai Mental Health Center
Model: Parallel | Masking: None
Other Study IDs: 2006L01603; SMHC-106
Record Dates: First submitted 2009-07-05; First posted 2009-07-07 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: duloxetine; pharmacokinetics; antidepressant; antidepressive agents; depression; psychotropic drugs; safety; Chinese; HAN; BDNF
MeSH Terms: conditions — Depression | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- low dose group (Experimental): single oral administer 15mg duloxetine
  Interventions: Drug: duloxetine
- moderate dose group/multiple dose group (Experimental): single oral duloxetine 30mg, after that repeat 7 oral duloxetine 30mg/d
  Interventions: Drug: duloxetine
- high dose group/crossover group (Experimental): single oral duloxetine 60mg, after that single oral innovator duloxetine 60mg
  Interventions: Drug: duloxetine

INTERVENTIONS:
Drug: duloxetine — 30mg, oral administer; step 1: single dose; step 2: multiple dose, 7 days
  Other Names: Generic duloxetine
  Arms: moderate dose group/multiple dose group
Drug: duloxetine — 15mg, oral administer
  Other Names: generic duloxetine
  Arms: low dose group
Drug: duloxetine — 60mg, oral administer; step 1: generic duloxetine; step 2: Innovator duloxetine
  Other Names: generic duloxetine; innovator duloxetine
  Arms: high dose group/crossover group

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics of duloxetine hydrochloride tablets in Chinese Han Healthy Subjects. The single oral dose and multiple oral dose of the drug in the body and the effects of different dosages of the drug will also be evaluated.

DETAILED DESCRIPTION:
This is an open, parallel assignment (low-dose, moderate-dose and high-dose), inpatient, sequential-group pharmacokinetics study of single oral administered and multiple oral administered to healthy Chinese male and female subjects at a single investigational site. All subjects are from the Chinese Han race.

Approximately 36 healthy male and female Chinese subjects will participate in this study. One half of the subjects enrolled in each dose group will be female. Twelve subjects will be enrolled in each of 3 dose level groups.

Safety will be evaluated from self-reported adverse events, scheduled physical examination, vital signs, 12-lead ECGs, and clinical laboratory test results.

Single-dose blood samples (5 mL) will be obtained within 2 hours before test article administration and at 1, 2, 3, 4, 5, 6, 8, 12, 15, 24, 36, 48, and 72 hours after test article administration.

Multiple-dose (subjects of moderate dose group finished first step single-dose 30mg trial, one week later, will be repeatedly administered duloxetine 30 mg 7days) blood samples (5 mL) will be obtained at 4th, 5th, 6th and 7th day before test article administration (to test the valley concentration)and at 1, 2, 3, 4, 5, 6, 8, 12, 15, 24, 36, 48, and 72 hours after last test article administration (7th day).

Cross-over (subjects of high dose group finished first step single-dose 60 mg generic duloxetine trial, one week later, will be administered single-dose innovator duloxetine 60 mg) blood samples will be obtained as same as first step.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese Han male or female determined by the investigator on the basis of medical history and physical examination
* Age from 18 to 45 years old at screening
* Body mass index (BMI) from 19~24 kg/m2 and body weight ≥ 50 kg at screening
* Normal clinical laboratory test results or 'no clinical significantly abnormal' results judged by the investigator at screening
* Subjects can comply with all requirements of the study according to study procedure
* A sighed and dated ICF (informed consent form) with approval by IEC

Exclusion Criteria:

* Participation in any drug trial within 1 month prior to enrollment into this study
* Known hypersensitivity to duloxetine hydrochloride or relative compounds
* Abnormal 12-lead electrocardiogram (ECG) results and increasing risk to participate this study determined by investigator
* Presence or history of any medical disorder, including cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, psychiatric and neurologic system, or medical conditions that would significantly affect the absorption, distribution, metabolism, or excretion of investigational drug, or increase risk to administer investigational drug, or interfere explanation for data
* History of hepatitis B and/or HBsAg (+)
* Serum HIV antibody (+) or hepatitis C Antibody (+)
* Female subjects of childbearing potential with a positive human chorionic gonadotropin (HCG) test or lack of a reliable method of contraception
* History of blood donor within 3 months prior to enrollment
* History of drug abuse or alcoholism
* Use any drugs including traditional Chinese Medicine within 1 week prior to enrollment
* Any unsuitable subjects judged by the investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics as evaluated from blood concentrations of duloxetine | 2 months

SECONDARY OUTCOMES:
Safety and tolerability as evaluated from reported adverse events, scheduled physical examinations, vital sign measurements, cardiac rhythm monitoring, 12 lead ECG and clinical laboratory results | 2 months
Serum BDNF level as evaluated from blood sample | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Huafang LI, MD, PhD, Principal Investigator — Drug Clinical Trial Office, Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China